CLINICAL TRIAL: NCT06224309
Title: A Phase 1/2 Study to Evaluate the in Vivo Biodistribution, Radiation Dosimetry and a Preliminary Assessment of the Diagnostic Performance of [18F]BL40
Brief Title: Preliminary Assessment of [18F]BL40 in PET/CT Scans
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H23-03813
Record Dates: First submitted 2023-12-27; First posted 2024-01-25 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Diffuse Large B-cell Lymphoma; Multiple Myeloma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Chronic Lymphocytic Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Multiple Myeloma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 18F-BL40 PET/CT scan: Each subject will have two PET/CT scans, one using 18F-BL40 and the other using 18F-FDG. The 18F-BL40 radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada. 18F-FDG is considered standard care and has been approved by Health Canada.
  Interventions: Diagnostic Test: 18F-BL40 PET/CT; Diagnostic Test: 18F-FDG PET/CT; Diagnostic Test: Routine Blood Draw - Phase 1 only

INTERVENTIONS:
Diagnostic Test: 18F-BL40 PET/CT — Vital signs will be recorded prior to the BL40 injection. Each study subject will have an intravenous catheter inserted. Prior to the radiotracer injection an ultra low dose CT will be taken. Subjects are positioned supine, arms down. The subject will receive a bolus intravenous dose of the 18F-BL40 from an approved study supplier site. A Dynamic PET scan will be taken of the heart. Then a serial whole body PET scan will be done. Vital signs will be taken again and the subject will have a bathroom break. The patient will return to the scanner bed for a standard low dose CT and whole body PET scan. Vital signs will be taken again, and subject will be allowed to use the washroom again. The subject will return to the scanner bed for the final time for an ultra low dose CT and whole body PET scan. A final set of vitals will be taken and the subject will be discharged.
Diagnostic Test: 18F-FDG PET/CT — The patient will return on another day for the 18F-FDG PET/CT scan. A fasting period of 6 hours is required before this scan.
  Each study subject will have an intravenous catheter inserted. The subject will receive a bolus intravenous dose of the radiotracer from an approved study supplier site.
  The subject will rest in a comfortable chair for 60 minutes. The subjects will then be taken to a designated washroom and asked to void prior to being scanned in order to clear excreted radiotracer activity from the urinary tract.
  Subjects are positioned supine, arms down, and centered on the scanner bed and the PET/CT images will be acquired.
Diagnostic Test: Routine Blood Draw - Phase 1 only — Complete blood counts and routine clinical chemistry performed before and repeated within 18-72 hours after 18F-BL40 administration.

SUMMARY:
CXCR4 is type of receptor that has been detected in more than twenty different subtypes of cancers. Most of these cancers are associated with negative symptoms that worsen over time resulting in great disability and poor function. There is a need for novel tracers to image CXCR4-expressing tumors for better detection, staging, and monitoring of aggressive cancers without the need for invasive biopsy procedures that may not always properly capture the extent of a patient's disease.

This study looks to assess the safety and efficacy of a novel radiopharmaceutical known as 18F-BL40 through its use in a PET/CT scan. Participants will receive 2 PET/CT scans:

18F-BL40 and 18F-FDG as part of this study.

DETAILED DESCRIPTION:
This is a prospective registry study to evaluate the diagnostic utility of 18F-BL40 PET/CT to stage patients with CXCR4-expressing tumors, localize sites of tumors and assess safety and biodistribution of this drug in PET/CT scans.

Each subject will receive two PET/CT scans, one using 18F-BL40 and the other using 18F-FDG. The 18F-BL40 radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada. 18F-FDG is considered standard care and has been approved by Health Canada.

Follow-up assessments: All subjects will be contacted by phone the day after the injection of 18F-BL40. The subjects will be asked if they experienced any undesirable effects during the 18-72 hours after the administration of 18F-BL40. The local site attending nuclear medicine physician will then make an assessment as to whether these effects are likely related to 18F-BL40 administration.

All subjects will be followed for at least 6 months following the 18F-BL40 PET/CT exam. The evaluation will include a chart review of available imaging, laboratory tests, and treatment. The data required can be obtained from a review of the patient's paper and electronic charts, supplemented by telephone contact as needed to complete the information.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years
2. Life expectancy ≥3 months
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Participants with newly diagnosed or documented recurrent malignancy with one of the following cancers:

   * Diffuse large B-Cell lymphoma
   * Multiple myeloma
   * Mantle cell lymphoma
   * Marginal zone lymphoma
   * Chronic lymphocytic leukemia/small cell lymphoma
   * Waldenström Macroglobulinemia
5. For all indications except multiple myeloma, the participants at the time of enrolment must either be at initial presentation with histologically confirmed lymphoma, or have the presence of measurable disease by computed tomography (CT) and/or magnetic resonance imaging (MRI) or at least one visualized lesion on positron emission tomography (PET)/CT imaging (from an [18F]FDG PET) within 60 days of enrolment. In the case of participants with multiple myeloma, there must be documented relapse or progressive disease by MRI or [18F]FDG PET/CT imaging, or measurable disease within 60 days of enrolment (serum M-protein ≥0.5 g/dL or urine Bence-Jones protein ≥200 mg/24 hours).

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Medically unstable (e.g., acute illness, unstable vital signs)
3. Unable to lie supine for the duration of imaging
4. Unable to provide written consent
5. Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm)
6. Participants with widespread liver metastases occupying more than 50% of the liver volume will not be eligible to participate in this study as this would preclude assessment of normal liver activity for dosimetry purposes.
7. Participants who have received chemotherapy or dexamethasone (> 4 mg/day) within 3 weeks or antibody therapy within 6 weeks prior to the [18F]BL40 or [18F]FDG PET/CT scans.
8. Participants who have received radiotherapy in the previous 6 weeks prior to [18F]BL40 or [18F]FDG PET/CT scans to sites of measurable active disease.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective, open-label trial in patients with newly diagnosed or documented recurrent malignancy with one of the following cancers:
  * Diffuse large B-Cell lymphoma
  * Multiple myeloma
  * Mantle cell lymphoma
  * Marginal zone lymphoma
  * Chronic lymphocytic leukemia/small cell lymphoma
  * Waldenström Macroglobulinemia
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To determine the tolerability of [18F]BL40 | 1 hour post injection, 2 hours post injection and 18-72 hours post injection
  Occurrence of dose-limiting toxicities (DLTs) per protocol.
To determine the Absorbed doses (ADs) to normal organs and tumors per unit of administered activity of [18F]BL40 | 6 months
  Absorbed doses (ADs) to organs and tumors per unit of administered activity is measured in units Gy/MBq.
  (Tumor, individual organ dose and whole-body effective dose)
To evaluate the proportion of participants with tumors shown by [18F]BL40 PET/CT | 1 year
  Proportion of patients with [18F]BL40 positive disease at core reading.
To determine Time Integrated Activity Coefficients for organ and tumor for [18F]BL40 | 6 months
  Average time the activity spends in the organ or tumor, measured in units MBq·h/MBq
To determine the safety of [18F]BL40 | 1 hour post injection, 2 hours post injection and 18-72 hours post injection
  Proportion of subjects with adverse events (AEs), Grade 3 or above AEs, drug-related AEs

SECONDARY OUTCOMES:
The proportion of patients in whom [18F]BL40 and [18F]FDG detect disease | 1 year
  The proportion of patients in whom one or more target lesions are detected by the core readers
To compare the number of lesions identified in [18F]BL40 and [18F]FDG | 1 year
  Scan features for comparison may include, but are not limited to:
  Total number of lesions detected
To assess tumour detectability and image quality by means of standardised uptake values (SUV) for tumour lesions in [18F]BL40 compared to 2[18F]FDG PET/CT (SUVmax, SUVpeak, tumour to background ratio for liver, blood, and lung, contrast to noise ratio) | 1 year
  Standard Uptake Values (SUV)
  mean SUV
  maximum SUV
  peak SUV
  Tumor tissue to Background tissue ratio, Tumor/blood; Tumor/Liver; Tumor/ kidney
To compare the lesions identified in [18F]BL40 and [18F]FDG | 1 year
  Scan features for comparison may include, but are not limited to:
  Site of lesions
To assess reader confidence | 1 year
  Diagnostic confidence on a three-point scale (high, moderate and low)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Alberts, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No